CLINICAL TRIAL: NCT02386254
Title: Adaptation of a Premorbid Function Scoring System as a Predictor for Intensive Care Unit Mortality
Acronym: ECOG
Status: Withdrawn | Type: Observational
Why Stopped: The study was administratively inactivated by the IRB after the PI did not submit the annual review and did not respond to the IRB's expiration letters.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: ECOG 9058
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: ICU Mortality; ICU Morbidity
Keywords: premorbid; scoring system; ECOG; ICU; morbidity; mortality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate whether a premorbid functioning scoring system such as the ECOG system can be adapted to predict ICU morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years and older admitted to the Presbyterian Hospital intensive care units under the medical ICU service.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the critical care units of Presbyterian Hospital under the care of the medical ICU service with any diagnosis will be assessed for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Mortality | 30-day
  Data will be expressed as mean + SD. Non parametric data will be expressed as median with interquartiles. Student t-test will be used to compare the normally distributed data, and the Mann-Whitney U test will be used for non parametric data. Chi-Squared test will be used to assess for trend between the ECOG score and the 30-day mortality. The investigators will use logistic regression analysis to determine the factors (including the ECOG score) associated with the 30-day mortality. Significance will be accepted for p values < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Kellie Jones, MD, Principal Investigator — Faculty
Locations (1):
- OU Medical Center, Oklahoma City, Oklahoma, United States